CLINICAL TRIAL: NCT04997512
Title: FreeSTyle LibRe and hospitAl Admissions, morTality and qUality of Life in High Risk Type 2 diabeteS Patients
Brief Title: Freestyle Libre and Hospital Admissions in Type 2 Diabetes
Acronym: STRATUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Collaborators: Abbott Diabetes Care (Industry)
Responsible Party: Principal Investigator, Ramzi Ajjan, Professor of metabolic medicine, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRATUS
Record Dates: First submitted 2021-07-26; First posted 2021-08-09 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes
Keywords: Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial (not blinded due to study design)
Masking Description: Unable to mask participants and trailists due to study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): Participants are returned to the care of their usual diabetes care provider following randomisation. They will donate blood and urine samples as well as completing diabetes specific questionnaires at 0 and 6 months. They will also wear a blinded glucose sensor (freestyle Libre PRO) for a two week period at month 6.
- Intervention arm (Experimental): Participants will be randomised at baseline. They will provide blood and urine samples at months 0 and 6 as well as fill in diabetes specific questionnaires. They will receive education surrounding hypoglycaemia at baseline from a diabetes specialist nurse. They will wear a freestyle libre device which is changed every two weeks for a period of 6 months. At weeks 2,4,12 and 24 they will have their diabetes medication adjusted by the diabetes specialist nurse/diabetes doctor according to their blood glucose profiles, analysed from the data generated by freestyle libre.
  Interventions: Device: Freestyle libre; Other: Nurse led structured intervention - hypoglycaemia education and diabetes treatment modification modification

INTERVENTIONS:
Device: Freestyle libre — A glucose sensor (flash) which measures interstitial blood glucose every 15 minutes or on demand.
  Arms: Intervention arm
Other: Nurse led structured intervention - hypoglycaemia education and diabetes treatment modification modification — An education programme surrounding avoidance of hypoglycaemia at baseline. Regular review (weeks 2, 4, 12 and 24) and adjustment of diabetes medications based on freestyle libre data.
  Arms: Intervention arm

SUMMARY:
This study aims to investigate the utility of a combination of structured nurse led intervention and the use of Freestyle libre in adults with type 2 diabetes who have suffered an episode of severe hypoglycaemia in terms of mortality, unscheduled healthcare contacts and quality of life.

DETAILED DESCRIPTION:
It is increasingly recognised that hypoglycaemia carries risk to individuals with all forms of diabetes. Research has shown high rate of mortality in those with type 2 diabetes following an episode of severe hypoglycaemia and a previous pilot trial conducted in the UK suggested that this could be improved by a structured nurse led intervention aimed at modifying glycemic therapy to avoid hypoglycaemia, instigating regular blood glucose monitoring and providing education to participants on common triggers for hypoglycaemia and how to avoid them.

In this trial, the investigators will randomise individuals with type 2 diabetes who have suffered an episode of severe hypoglycaemia requiring emergency service call out to two arms. One arm will receive standard of care/treatment as usual and the other will receive a structured nurse led intervention as well as the use of a flash glucose monitoring system, Freestyle libre.

Active participation in the trial for both arms will be a total of twelve months (with the main intervention months 0-6.) Participants electronic records will be analysed for death and unscheduled healthcare contacts for a total of two years after recruitment.

The primary outcome measure is mortality between groups. Secondary outcomes include the use of estimated HbA1c (a variable produced by the freestyle libre device) compared to laboratory HbA1c, quality of life measures, effects on glycemic control and the number of unscheduled healthcare contacts.

ELIGIBILITY:
Inclusion criteria

* Aged >18
* Confirmed diagnosis of type 2 diabetes
* Suffered an episode of severe hypoglycaemia requiring ambulance call out
* Able to provide informed written consent

Exclusion criteria

* A form of diabetes mellitus which is not type 2 or the diagnosis is uncertain
* Currently pregnant
* Dialysis dependent renal failure
* Unable to provide informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality at 2 years | 2 years
  Rates of death between groups at 2 years

SECONDARY OUTCOMES:
All-cause mortality at 1 year | 12 months
  Mortality at 12 months from randomisation
Cardiovascular mortality at 1 year | 1 year
  Mortality from a cardiovascular cause at 1 year
Cardiovascular mortality at 2 years | 2 years
  Mortality from a cardiovascular cause at 2 years
Number of unscheduled healthcare contacts | 2 years after randomisation
  Number of unscheduled healthcare contacts (emergency services, hospital attendances, primary care attendances) 1 year prior to randomisation and 2 years after
Comparison between estimated HbA1c and laboratory HbA1c | 6 months
  A comparison between estimated HbA1c (freestyle libre generated) and laboratory HbA1c values across the whole study cohort at 0 and 6 months
Change from baseline in HbA1c | 6 months
  Change from baseline HbA1c at 6 months between both groups
Scores from Diabetes distress scale | Tested at 0 and 6 months
  A questionnaire which assessed the emotional burden diabetes has on the participant. 4 different domains are tested across 17 questions. An overall score is calculated (each question is ranked 1-6 by participants) and the total score is divided by 17. The higher the score (1-6) the more diabetes distress the participant is under. Scores are also calculated across each domain. These are 1) emotional burden 2) Physician associated distress 3) regimen associated distress 4) interpersonal distress
Scores from diabetes quality of life scale (DQOL) | Tested at 0 and 6 months
  This is a questionnaire with 15 questions filled in by participants. Each question is ranked 1-5 with a score of 5 conveying the worst score. Scores therefore range from 15 to 75 with a score of 75 indicating very poor quality of life as a result of diabetes and 15 very good.
Scores from treatment satisfaction scale (DTSQc) | Tested at 0 and 6 months
  This is a questionnaire assessing participant satisfaction with the treatment of their diabetes. It comprises 8 questions with each scored from 3 to negative 3. A score of 3 on a question indicates very good satisfaction whereas negative 3 that the participant is most dissatisfied. Therefore a maximum score of 24 is possible with a low score of negative 24. The higher the score, the more satisfied the participant is with their diabetes treatment.
Scores from GOLD score | Tested at 0 and 6 months
  A 1-7 scale which asks participants how likely they are to recognise hypoglycaemia. 7 indicates they have severe hypoglycaemia awareness and 1 that they are fully hypoglycaemic aware. Therefore the higher the score, the more hypoglycaemic unawareness the participant perceives themself as having.

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi A Ajjan, PHD, Principal Investigator — University of Leeds
Locations (1):
- Diabetes centre, St James hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be available on reasonable request to the investigators

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04997512/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT04997512/ICF_001.pdf